CLINICAL TRIAL: NCT05716581
Title: The Identification of Prognostic Factors for Patients Undergoing Ablation for Atrial Fibrillation
Brief Title: Prognostic Factors for Ablation of Atrial Fibrillation
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: Prognostic AF
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Spectral Analysis; Vectorcardiography; Heart Rate Variability
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Catheter ablation — Catheter ablation for atrial fibrillation will be done according to the current medical praxis. Pulmonary vein isolation using either radiofrequency or pulsed-field ablation will be done in all patients. In patients with non-paroxysmal AF, additional ablation lesions (posterior wall ablation, roof or mitral isthmus line, ablation of complex fractionated atrial electrograms) could be done based on the operator´s discretion

SUMMARY:
The aim of the study is to find factors associated with sinus rhythm maintenance after catheter ablation for atrial fibrillation.

DETAILED DESCRIPTION:
Catheter ablation presents the most effective kind of treatment for atrial fibrillation (AF). However, its efficacy is still limited, and AF reoccurs in approx. 30% of patients during the first year after ablation.

Several factors associated with AF recurrences were found, such as dilated left atrium, higher age, or the duration of AF before the ablation. As it was shown, the detailed analysis of the ECG before the ablation could also serve several important factors that could predict AF reoccurrence.

In the study, all participants who will be referred for AF ablation in the study center will be enrolled. Pre-procedural ECG on the day of the ablation (just during the procedure) will be analysed using several methods: 1) spectral analysis (dominant AF frequency will be determined), 2) heart rate variability (for time and frequency domain analysis), 3) vectorcardiography. All ECG recordings will be analyzed using matlab software.

All participants will have regular follow-up checks at 3, 6, and 12 months after ablation including 24-hour Holter recordings. Based on the rhythm presence during the follow-up, participants will be divided in two groups: 1) AF group (patients with AF recurrences) and 2) sinus rhythm (SR) group (patients without AF reoccurrence during follow-up). AF reoccurrence will be determined at a presence of AF or any other atrial tachycardia lasting > 30 sec. The results of pre-procedural ECG analysis will be compared between both groups. Logistic regression will be done to determine optimal combination of parameters associated with AF freedom.

ELIGIBILITY:
Inclusion Criteria:

* atrial fibrillation

Exclusion Criteria:

* absent of informed content

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients indicated for the catheter ablation for atrial fibrillation in our center will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
AF reoccurrence during follow-up | 1 year after the ablation
  AF freedom will be defined as freedom from atrial fibrillation or any other regular atrial tachycardia lasting > 30sec. Rhythm monitoring will be done using regular Holter recordings

IPD SHARING:
Plan to Share IPD: Yes
AFter study completion, data will be available on the request.
Time Frame: After study completion